CLINICAL TRIAL: NCT00068666
Title: A Systemic Temozolomide Treatment Of Melanoma Present In The Central Nervous System
Brief Title: Temozolomide and Radiation Therapy in Treating Patients With Stage IV Malignant Melanoma With Measurable and Unresectable Cancer of the Central Nervous System
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N0274; CDR0000327811 (Registry Identifier: PDQ (Physician Data Query)); NCI-2012-02554 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Melanoma (Skin); Metastatic Cancer
Keywords: stage IV melanoma; recurrent melanoma; tumors metastatic to brain
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Brain Neoplasms | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- radiation + temozolomide (Experimental): Patients receive concurrent chemoradiotherapy comprising whole brain radiotherapy daily on days 1-5, 8-13, and 16-21 and oral temozolomide daily on days 1-5. Subsequent treatment with temozolomide repeats every 4 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 2 months.
  Interventions: Drug: temozolomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: temozolomide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining temozolomide with radiation therapy may make the tumor cells more sensitive to radiation therapy and kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving temozolomide together with radiation therapy works in treating patients with stage IV malignant melanoma with measurable and unresectable cancer limited to the central nervous system.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with stage IV malignant melanoma with measurable and unresectable disease of the central nervous system treated with temozolomide and radiotherapy.

Secondary

* Determine the safety of this regimen in these patients.
* Determine the survival of patients treated with this regimen.
* Determine the effect of this regimen on performance status and mental status of these patients.
* Determine the response of extra-cranial disease in patients treated with this regimen.

OUTLINE: Patients receive concurrent chemoradiotherapy comprising whole brain radiotherapy daily on days 1-5, 8-13, and 16-21 and oral temozolomide daily on days 1-5. Subsequent treatment with temozolomide repeats every 4 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A total of 18-41 patients will be accrued for this study within 13-30 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV malignant melanoma with measurable and unresectable disease limited to the central nervous system (CNS)

  * Study entry within 14 days of diagnosis of brain metastases
* Recursive partitioning analysis class I or II
* Disease for which no known standard therapy exists that is potentially curative or proven capable of extending life expectancy
* No meningeal carcinomatosis based on imaging studies or on positive results from CSF analysis
* No evidence of metastatic disease outside of the CNS

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic

* AST no greater than 3 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 3 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent uncontrolled infection
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer treated with local resection only
* No prior allergy or intolerance to dacarbazine
* No hypersensitivity to temozolomide or any of its components

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biologic therapy
* More than 4 weeks since prior immunotherapy

Chemotherapy

* No prior temozolomide
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered

Endocrine therapy

* Concurrent steroids allowed if dose stable for at least 7 days prior to CNS imaging

Radiotherapy

* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 15% of the bone marrow
* No prior radiotherapy to the head and neck area
* No prior radiosurgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-01; Primary Completion 2005-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Confirmed response rate | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival | Up to 5 years
Overall survival | Up to 5 years
Change in performance status | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (45):
- United States (45):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Grandview Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Result] Schild SE, Behl D, Markovic SN, Brown PD, Sande JR, Deming RL, Rowland KM Jr, Bearden JD. Brain metastases from melanoma: is there a role for concurrent temozolomide in addition to whole brain radiation therapy? Am J Clin Oncol. 2010 Dec;33(6):633-6. doi: 10.1097/COC.0b013e3181c4c54b. PMID 20042969